CLINICAL TRIAL: NCT00583167
Title: CNS Viral Dynamics and Cellular Immunity During AIDS
Brief Title: CNS (Central Nervous System) Viral Dynamics and Cellular Immunity During AIDS
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, David Haas, Professor of Medicine, Vanderbilt University
Other Study IDs: 050001; R01MH071205 (NIH)
Record Dates: First submitted 2007-12-26; First posted 2007-12-31 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; CNS; brain; affects
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, plasma, CSF
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- A1: HIV-infected subjects who are at least 18 years of age, with no ART in the previous 3 months, and with plasma HIV-1 RNA >20,000 copies/mL. CD4+ T cell count >200 cells/mm3. Group A1 will undergo continuous CSF ( cerebrospinal fluid) sampling via intrathecal catheter.
- A2: HIV-infected subjects who are at least 18 years of age, with no ART in the previous 3 months, and with plasma HIV-1 RNA >20,000 copies/mL. CD4+ T cell count <200 cells/mm3. Group A2 will undergo continuous CSF sampling via intrathecal catheter.
- B: HIV-infected subjects who are at least 18 years of age, with no ART in the previous 3 months, and with plasma HIV-1 RNA >20,000 copies/mL. Group B will not undergo continuous CSF sampling, but will undergo sparse CSF sampling by lumbar punctures.

SUMMARY:
Understanding whether or not viral replication occurs in the brain during chronic untreated HIV-1 infection is of undeniable importance, and has implications for treatment and research priorities. Evidence suggests that viral replication in the CNS occurs at the extremes of HIV-1 disease. Brain involvement has been reported during acute infection, and there is convincing evidence of CNS viral replication during HIV-associated dementia (HAD) and advanced AIDS. Some human and primate data suggest that viral RNA and proteins may be absent from brains of some individuals with chronic untreated HIV-1 infection despite abundant proviral DNA. However, the extent of viral replication in the brain is not known for most of the 42 million people worldwide living with untreated HIV-1 infection.

Why is viral replication in the brain such a pivotal issue? Microglial cells and macrophages are primary targets for intrathecal HIV-1 replication, and this can promote neuronal injury through direct effects of gp120 and tat, and indirect induction of toxic mediators. Low-grade injury over years or decades would likely be deleterious, particularly as the population ages. Because treatment guidelines allow systemic HIV-1 replication to continue until CD4+ T cell counts decline considerably, antiretroviral therapy (ART) is not recommended for many persons living with HIV. Demonstrating replication in the brain during chronic HIV-1 infection may affect treatment strategies and encourage investigation.

Identifying factors that modulate intrathecal viral replication is equally important. Anti-HIV-1 cytotoxic T lymphocytes (CTL) partially control systemic viral replication and delay disease progression. Although available data has been provocative, the role of anti-HIV CTL in the CNS has received little attention. To fill this gap we will examine relationships between intrathecal viral replication, CTL responses, and glial activation/proliferation during HIV-1 infection. These studies will be relevant not only to AIDS but to other inflammatory diseases of the CNS as well.

ELIGIBILITY:
Inclusion Criteria:

* (All subjects in Groups A1, A2 and B):
* At least 18 years of age.
* No more than one month of ART in the past.
* No ART in the previous 3 months.
* Platelet count >100,000 cells/mm3 on most recent determination within 60 days prior to first study lumbar puncture.
* Normal prothrombin time (PT) and partial thromboplastin time (PTT) on most recent determination within 60 days prior to first study lumbar puncture.
* Among individuals with past ART experience, the ability to construct an ART regimen predicted to completely suppress plasma HIV-1 RNA, based on results of viral susceptibility testing that is done as a routine part of clinical practice.
* Plasma HIV-1 RNA >20,000 copies/mL.
* Additional Inclusion Criteria for Groups A1 and A2.
* Group A1:
* CD4+ T cell count >200 cells/mm3.
* CSF HIV-1 RNA >2,000 copies/mL on screening lumbar puncture.
* No history of significant allergy to beta lactam antibiotics, including penicillins and cephalosporins.
* No history of allergy to vancomycin.
* Group A2:
* CD4+ T cell count <200 cells/mm3.
* CSF HIV-1 RNA >2,000 copies/mL on screening lumbar puncture.
* No history of significant allergy to beta lactam antibiotics, including penicillins and cephalosporins.
* No history of allergy to vancomycin.

Exclusion Criteria:

* Evidence of CNS opportunistic infections or space occupying lesion.
* History of significant CNS disorder unrelated to HIV infection such as trauma, congenital malformations or genetic disorders.
* History of seizures.
* As determined by the investigator, a significant active or previous history of cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, or endocrine disease(s) that would interfere with study participation.
* Evidence or suspicion of vascular or Alzheimer's type dementias.
* Evidence or suspicion of Parkinson's disease.
* History of allergy to lidocaine.
* Implanted metal objects that make MRI contraindicated. This may require consultation with colleagues in the Vanderbilt Dept. of Radiology.
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment or prior to study drug administration.
* Women of childbearing potential (WOCBP) who are unwilling or unable to use an adequate method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected subjects who are at least 18 years of age, with no ART in the previous 3 months, and with plasma HIV-1 RNA >20,000 copies/mL. Individuals with past ART experience must have the ability to construct an ART regimen predicted to completely suppress plasma HIV-1 RNA, based on results of viral susceptibility testing that is done as a routine part of clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2006-03; Primary Completion 2009-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To characterize intrathecal viral replication during chronic untreated HIV-1 infection, and to assess how intrathecal viral replication relates to stage of HIV-1 disease. | end of study
To measure intrathecal and systemic cellular immune responses against HIV-1 and to assess how these responses relate to intrathecal viral replication. | end of study
To correlate intrathecal viral replication and anti-HIV CTL responses with the degree of glial activation/proliferation and neuronal dropout in the brain. | end of study

CONTACTS AND LOCATIONS:
Overall Officials: David W. Haas, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt AIDS Clinical Trials Center, Nashville, Tennessee, United States